CLINICAL TRIAL: NCT00308464
Title: A Double Blind Parallel Group Randomised Multiple Dose Study To Evaluate The Pharmacodynamic Response And Safety Of PHA-794428 In Adult Growth Hormone Deficient Patients
Brief Title: A Study To Evaluate The Dose Response And Safety Of PHA-794428 In Adults With Growth Hormone Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6391003
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

INTERVENTIONS:
Drug: PHA-794428

SUMMARY:
The purpose of this study is to explore the safety, toleration and dose response of PHA-794428 after multiple weekly injections in male and female growth hormone deficient patients.

DETAILED DESCRIPTION:
The study terminated on 10-Dec-2007. Pfizer's decision to terminate the program was due to cases of injection-site lipoatrophy that were reported in the clinical Phase 2 studies after a single injection of PHA 794428.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with severe AGHD.
* Hypopituitary patients must be on adequate hormone replacement therapy for at least 6 months.

Exclusion Criteria:

* AGHD patients with uncontrolled pituitary tumor growth.
* Tumors within 3 mm of the optic chiasm.
* Patients with diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Responder status at visits 9 (week 4) and 14 (week 7), where responder is defined as a patient who has achieved an IGF-1 level above the mid-point of the age-related normal range.

SECONDARY OUTCOMES:
Change in PD and glycemic control | At weeks 4 and 7
Change in PK concentrations.
ALT, AST greater than 3.0 times ULN at any visit
Anti-hGH and anti PHA-794428 antibody production
Change in body weight | At week 4 and follow-up
Injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Belgium (3):
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
- Czechia (2):
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Prague
- Denmark (4):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Koebenhavn OE
  - Pfizer Investigational Site, Odense C
- France (3):
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Reims
- Germany (3):
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, München
- Italy (5):
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Torino
- Pfizer Investigational Site, Leiden, Netherlands
- Poland (2):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Wroclaw
- Slovakia (2):
  - Pfizer Investigational Site, Ľubochňa, Slovakia
  - Pfizer Investigational Site, Bratislava
- Spain (3):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Granada, Granada
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
- Sweden (4):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Umeå
- United Kingdom (3):
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Oxford

REFERENCES:
- [Derived] Touraine P, D'Souza GA, Kourides I, Abs R, Barclay P, Xie R, Pico A, Torres-Vela E, Ekman B; GH Lipoatrophy Study Group. Lipoatrophy in GH deficient patients treated with a long-acting pegylated GH. Eur J Endocrinol. 2009 Oct;161(4):533-40. doi: 10.1530/EJE-09-0422. Epub 2009 Aug 4. PMID 19654233
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6391003&StudyName=A%20Study%20To%20Evaluate%20The%20Dose%20Response%20And%20Safety%20Of%20PHA-794428%20In%20Adults%20With%20Growth%20Hormone%20Deficiency